CLINICAL TRIAL: NCT01909960
Title: Benefit of Flow Magnetic Resonance Imaging in the Management of Normal Pressure Hydrocephalus
Brief Title: Flow MRI in Normal Pressure Hydrocephalus
Acronym: HydroFlux
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PHRCIR11-DR-BALEDENT; 2011-A01633-38 (Registry Identifier: RCB)
Record Dates: First submitted 2013-05-24; First posted 2013-07-29 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Normal Pressure Hydrocephalus
Keywords: Normal pressure hydrocephalus; Flow MRI; Dementia; Cerebrospinal fluid; Shunt
MeSH Terms: conditions — Hydrocephalus, Normal Pressure; Dementia | interventions — Hydrodynamics; Cerebrovascular Circulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgery (Experimental): Patients who will undergo flow imaging and neurosurgery (shunting). (25% of the studied population)
  Interventions: Other: Flow imaging
- Clinical follow-up (Experimental): Patients who will undergo flow imaging but not surgery (75% of the studied population)
  Interventions: Other: Flow imaging

INTERVENTIONS:
Other: Flow imaging — Quantitative flow study was performed by 2D phase-contrast velocity-encoded cine MRI (repetition/echo time, 15/7 ms; field of view = 140 x 140 mm²; matrix size = 256 x 128, flip angle = 25 degrees,one excitation, slice thickness = 5 mm). Cerebrospinal fluid and blood flows are measured with a velocity-encoding value of 5-10 cm/s and 80 cm/s respectively. Peripheral gating was used to cover the entire cardiac cycle with retrospective cardiac synchronization of 32 quantitative flow-encoded images per cycle.
  Clinical examination consists in Larson's score and MMSE
  Other Names: Flow MRI; Cine phase-constrast magnetic resonance imaging; CSF pulsatility; Hydrodynamic; Cerebral blood flow

SUMMARY:
Normal pressure hydrocephalus diagnosis based on quantitative study of cerebro-spinal fluid and blood flow by phase contrast magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* Ventricular dilation seen on morphological magnetic resonance imaging (MRI)
* Walking disorder
* Cognitive disorder
* Participants gave their written informed consent

Exclusion Criteria:

* Contra-indication to MRI
* Obstructive tumoral hydrocephalus
* Curatorship or tutorship
* Pregnancy or lactation
* No social assurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2012-05-03 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
cerebrospinal fluid (CSF) stroke volume evolution other 6 months | Day 1 (baseline), Day 180
  Measurement of cerebrospinal fluid (CSF) stroke volume via flow MRI at the Sylvius' aqueduct, pontine cistern and spinal spaces levels and determination of its evolution

SECONDARY OUTCOMES:
Blood flow analysis : evolution other 6 months | Day 1 (baseline), Day 180
  Assessment of arterial (internal carotids and cerebral arteries) and venous (sagittal sinus, straight sinus) blood flow in terms of mean cerebral blood outflow and stroke volume and determination of blood flow evolution.
Larson's score evolution over 6 months | Day 1, Day 180
  Record symptoms on walking, living conditions and urinary disorders
Neuropsychological test evolution over 6 months | Day1, Day 180
  Consists in mini mental status evaluation (MMSE) for cognitive evaluation
Blood flow analysis : evolution other one year | Day 1 (baseline) and Day 365
  Assessment of arterial (internal carotids and cerebral arteries) and venous (sagittal sinus, straight sinus) blood flow in terms of mean cerebral blood outflow and stroke volume and determination of blood flow evolution.
Larson's score evolution over one year | Day 1 and Day 365
  Record symptoms on walking, living conditions and urinary disorders
Neuropsychological test evolution over one year | Day1, Day 365
  Consists in mini mental status evaluation (MMSE) for cognitive evaluation
cerebrospinal fluid (CSF) stroke volume evolution other one year | Day1 (baseline), Day 365
  Measurement of cerebrospinal fluid (CSF) stroke volume via flow MRI at the Sylvius' aqueduct, pontine cistern and spinal spaces levels and determination of its evolution

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Balédent, PhD, Principal Investigator — CHU Amiens
Locations (2):
- France (2):
  - CHU Lille, Lille, Hauts-de-France
  - CHU Amiens, Amiens, Picardie